CLINICAL TRIAL: NCT01246479
Title: Long Term Immunity and Safety Following Vaccination With the Japanese Encephalitis Vaccine IC51(IXIARO®, JESPECT®) In a Pediatric Population in Non Endemic Countries. Uncontrolled, Phase 3 Follow-up Study
Brief Title: Long Term Immunity and Safety Following Vaccination With the JEV IC51 (IXIARO®, JESPECT®) in Pediatric Population In Non Endemic Countries. Uncontrolled, Ph3 FU-Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IC51-324
Record Dates: First submitted 2010-10-06; First posted 2010-11-23 (Estimated); Results first posted 2015-04-29 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- No treatment (Other): subjects will be followed up on immunity (analysis of blood samples) and safety
  Interventions: Procedure: Blood draw; Biological: IC51 has given in the parent study IC51-322

INTERVENTIONS:
Procedure: Blood draw — blood draw at Month 12, Month 24 and Month 36.
Biological: IC51 has given in the parent study IC51-322 — No more vaccinations in IC51-324 since this a study for long-term follow-up on safety and immunogenicity after vaccinations in parent study IC51-322.

SUMMARY:
The study investigates long-term immunity and safety of IC51 (IXIARO®, JESPECT®) in a pediatric population vaccinated in the parent study IC51-322.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have received two vaccinations in study IC51 322. (2) Subjects who were enrolled as part of the immunogenicity subgroup of study IC51-322.
* Male or female healthy subjects aged ≥ 9 months to < 21 years at the time of enrolment into this study.
* Written informed consent by the subject, the subject's legal representative(s), according to local requirements, and written informed assent of the subject, if applicable.

Exclusion Criteria:

* History of or clinical manifestation of any Flavivirus disease during study IC51-322.
* Vaccination against JE virus (JEV) (except with IC51) at any time prior or planned during this study.
* Participation in another study with an investigational product during study IC51-322 or IC51-324.
* History of or development of any immunodeficiency including post-organtransplantation after inclusion into study IC51-322.
* History of or development of an autoimmune disease during study IC51-322.
* Administration of chronic (defined as more than 14 days) immunosuppressants or other immune-modifying medications started during study IC51-322 up to first visit of study IC51-324. (For corticosteroids this means prednisone or equivalent at >= 0.05 mg/kg/day. Topical or inhaled steroids are allowed).
* Known infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV).
* Illicit drug use and/or a history of drug or alcohol addiction and/or current drug or alcohol addiction.
* Inability or unwillingness by the legal representative(s) and/or the subject (where applicable) to provide informed consent/assent and to abide by the requirements of the study.
* Persons who are committed to an institution (by virtue of an order issued either by the judicial or the administrative authorities).

Ages: 9 Months to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ayad, Dr., Study Chair — Valneva Austria GmbH
Locations (5):
- Tampa, Florida, United States
- Australia (2):
  - Brisbane
  - Melbourne
- Germany (2):
  - Berlin
  - Hamburg

REFERENCES:
- [Derived] Taucher C, Barnett ED, Cramer JP, Eder-Lingelbach S, Jelinek T, Kadlecek V, Kiermayr S, Mills DJ, Pandis D, Reiner D, Dubischar KL. Neutralizing antibody persistence in pediatric travelers from non-JE-endemic countries following vaccination with IXIARO(R) Japanese encephalitis vaccine: An uncontrolled, open-label phase 3 follow-up study. Travel Med Infect Dis. 2020 Mar-Apr;34:101616. doi: 10.1016/j.tmaid.2020.101616. Epub 2020 Mar 7. PMID 32156630

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Treatment
Started | 23
Completed | 18 (primary endpoint at Month 12)
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- No Treatment: subjects will be followed up on immunity (analysis of blood samples) and safety
  Blood draw: blood draw at Month 12, Month 24 and Month 36.
  IC51 was given in the parent study IC51-322: No more vaccinations in IC51-324 since this a study for long-term follow-up on safety and immunogenicity after vaccinations in parent study IC51-322.
Arm/Group | No Treatment
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Rate of Subjects With PRNT50 Titers of ≥ 1:10 at Month 12 After the First IC51 Vaccination (in Study IC51-322)
Description: Rate of subjects with PRNT50 titers of ≥ 1:10 at Month 12 after the first IC51 vaccination (in study IC51-322)
Time Frame: Month 12
Population: intention to treat population; assessment of seroprotection ~1 year post primary vaccination series in parent study IC51-322
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | No Treatment
Number analyzed (Participants) | 19
percentage of participants | 89.5 [68.6 to 97.1]

2. Secondary Outcome: GMT for JEV Neutralizing Antibodies Measured Using the PRNT at Month 12, 24 and 36 After the First IC51 Vaccination (in Study IC51-322)
Description: GMT for JEV neutralizing antibodies measured using the PRNT at Month 12, 24 and 36 after the first IC51 vaccination (in study IC51-322)
Time Frame: Month 12, 24 and 36
Population: Intent to Treat Population
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | No Treatment
Number analyzed (Participants) | 23
Titer
  Month 12 - Visit 2 | 47.8 [28.7 to 79.8]
  Month 24 - Visit 3: number analyzed (Participants) | 19
  Month 24 - Visit 3 | 75.4 [45.9 to 123.7]
  Month 36 - Visit 4 | 60.8 [34.8 to 106.1]

3. Secondary Outcome: Rate of Subjects With PRNT50 Titers of ≥ 1:10 at Months 24 and 36 After the First IC51 Vaccination (in Study IC51-322)
Description: Rate of subjects with PRNT50 titers of ≥ 1:10 at Months 24 and 36 after the first IC51 vaccination (in study IC51-322)
Time Frame: Month 24, 36
Population: Intent to Treat Population
Measure: Number; unit: percentage of participants
Arm/Group | No Treatment
Number analyzed (Participants) | 23
percentage of participants
  Seroprotection Rate - Month 24 - Visit 3: number analyzed (Participants) | 21
  Seroprotection Rate - Month 24 - Visit 3 | 91.3
  Seroprotection Rate - Month 36 - Visit 4: number analyzed (Participants) | 17
  Seroprotection Rate - Month 36 - Visit 4 | 89.5

4. Secondary Outcome: Rate of Subjects With SAEs Following Immunization up to Months 12, 24 and 36 After the First IC51 Vaccination (in Study IC51-322)
Description: Rate of subjects with SAEs following immunization up to Months 12, 24 and 36 after the first IC51 vaccination (in study IC51-322)
Time Frame: Months 12, 24 and 36
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | No Treatment
Number analyzed (Participants) | 23
Participants
  Month 12 - Visit 2 | 1
  Month 24 - Visit 3 | 2
  Month 36 - Visit 4 | 2

5. Secondary Outcome: Rate of Subjects With AEs and Medically Attended AEs up to Months 12, 24 and 36 After the First IC51 Vaccination (in Study IC51-322).
Description: Rate of subjects with AEs and medically attended AEs up to Months 12, 24 and 36 after the first IC51 vaccination (in study IC51-322).
Time Frame: Months 12, 24 and 36
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | No Treatment
Number analyzed (Participants) | 23
Participants
  Medically attended - Month 12 - Visit 2 | 7
  Medically attended - Month 24 - Visit 3 | 7
  Medically attended - Month 36 - Visit 4 | 7
  Any AE up to Month 12 | 8
  Any AE up to Month 24 | 8
  Any AE up to Month 36 | 8

ADVERSE EVENTS:
Time Frame: adverse event data were collected up to month 36 (i.e., approximately 3 years after primary immunization in the parent study IC51-322)
Arm/Group | No Treatment
Serious Adverse Events (participants affected / at risk) | 2/23
Other Adverse Events (participants affected / at risk) | 8/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Treatment (N=23)
Staphylococcal infection (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | No Treatment (N=23)
Otitis media acute (Infections and infestations) | 2
Pharyngitis streptococcal (Infections and infestations) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Skin papilloma (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days